CLINICAL TRIAL: NCT04252911
Title: Comparative Study Between Standard Vs Supralabial Bispectral Index Scores
Brief Title: Standard Vs Supralabial Bispectral Index Scores
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rajiv Gandhi Cancer Institute & Research Center, India (Other)
Responsible Party: Principal Investigator, Dr. Nitesh Goel, Consultant Anaesthesia, Principle investigator, Rajiv Gandhi Cancer Institute & Research Center, India
Other Study IDs: RajivGCIRC3
Record Dates: First submitted 2019-11-12; First posted 2020-02-05 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Intraoperative Awareness
Keywords: BIS; Intraoperative awareness
MeSH Terms: conditions — Intraoperative Awareness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Anaesthetised patients: 50 patients undergoing robotic surgeries under general anesthesia
  Interventions: Other: Bispectral index score

INTERVENTIONS:
Other: Bispectral index score — Bis value from two sites gives similar results
  Other Names: medtronic Bis Monitoring device

SUMMARY:
With the rise in number of surgeries, the medicolegal issues are on rise especially if patient had intraoperative awareness, which can also be detrimental to psychosocial behaviour of patient. Investigators plan to compare the BIS values, 'which is an indicator of awareness', from supralabial to standard forehead placement sites. If the results are corroborative then the supralabial site can be used for BIS monitoring in neurosurgical cases where it is not possible to to apply the forehead BIS strips.

DETAILED DESCRIPTION:
Consequences of intraoperative awareness could be hemodynamic disturbances, long-lasting psychological problem and medicolegal issues. Bispectral index (BIS) is the most widely used noninvasive method to estimate level of consciousness. Complex electroencephalography (EEG) parameter that converts raw EEG data from the frontal cortex into a single number between 100 (fully awake) and 0 (isoelectric EEG).

The BIS sensor is a single adhesive strip placed across the forehead. This position can be problematic in certain surgical procedures involving a neurosurgery, surgery involving fronto-temporal area of the face. Thus the need for alternative sites for BIS sensor placement is often felt. Several alternative sensor positions have been reported in literature like Occipital, Retroauricular, Mandibular. Each of these are found to have limitations. Investigators planned a study to compare the BIS values at two sites i.e. forehead(standard) versus supralabial placement of sensors so that BIS can be applied in neurosurgical cases if the two values relates statistically.

Sample size: Total of 50 patients will be recruited for the study. Every patient will act as control and test group as both standard forehead sensors and (test) supralabial sensors will be applied in same patient.

Method:

2 BIS sensors will be applied on each patient soon after the induction.

* Sensor 1: Frontal sensors will be applied with circle 1 at the center of the forehead; circle 2, 2.8 cm lateral to circle 1; and circle 3 on either temporal area between the corner of the eye and the hairline.
* Sensor 2: Supralabial sensors will be applied with circle 1 at the center of the upper lip at phrenulum, circle 4 adjacent to the lateral side of lip, and circle 3 at the ipsilateral temporal area.

Anaesthetic technique:

All patients will be given anti-aspiration prophylaxis with tab pantoperazole 20mg and tab. Granicetrone 2mg orally 2hrs before surgery with sips of water. After informed consent and recruitment as per inclusion-exclusion criteria, all patients will be premedicated with inj. midazolam mg. i.v. followed by intravenous induction with inj. propofol (1-2.5mg/Kg) along with Inj. Atracurium for muscle relaxation.

Intubation will be done after adequate muscle relaxation achieved in both groups. Intraoperatively muscle relaxation will be monitored by nerve stimulator. Aim will be to maintain BIS value of 40-60. Closed circuit anaesthesia along with inhalational gas flow rate of 1 litre/min will be maintained. Patient will be ventilated with oxygen and sevoflurane mixture along with propofol infusion @ 25-100 mcg/kg/min Patient will be reversed after monitoring TOF ratio once the surgery is over.

Monitoring: following 3 parameters

* BIS score
* Signal quality index (SQI)
* Electromyography (EMG) score

Data will be recorded at

* Before first surgical incision
* After the first surgical incision
* Every 15 minutes thereafter during the intraoperative period (maintenance)
* Pre extubation
* Post extubation (emergence).

Proposed Statistical Analysis:

The statistical analysis will be carried out using Statistical Package for Social Sciences (SPSS Inc.,IBM, version 24.0 for Windows).

Bland- Altman plot will be used to assess agreement between the values obtained from standard placement site and supralabial sensors

ELIGIBILITY:
Inclusion Criteria:

* Age group: 18-65 yrs
* ASA status: 1-3
* Use of endotracheal tube for securing the airway

Exclusion Criteria:

* Facial deformity : scars, cleft lip, mole etc
* Presence of beard and moustache
* Use of supraglottic device
* Patient under regional anaesthesia

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients of all genders of all age and BMI
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-01-20 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Intraoperative BIS values | from induction of anaesthesia till surgery is over upto 5 hours
  the values from both sites will be monitored

CONTACTS AND LOCATIONS:
Locations (1):
- Rajiv Gandhi Cancer Institute & Research Centre, New Delhi, National Capital Territory of Delhi, India